CLINICAL TRIAL: NCT00949832
Title: Vitamin D and Genetics in Nutritional Rickets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Jos University Teaching Hospital (Other)
Responsible Party: Thomas D. Thacher, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-006041
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Nutritional Rickets
Keywords: rickets; calcium; vitamin D; nutrition; child
MeSH Terms: conditions — Vitamin D Deficiency; Rickets | interventions — Vitamin D; Calcium; Ergocalciferols; Calcium Carbonate; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vitamin D + Calcium (Active Comparator): Vitamin D and calcium supplementation
  Interventions: Dietary Supplement: Vitamin D + Calcium
- Calcium (Placebo Comparator): Calcium supplementation
  Interventions: Dietary Supplement: Calcium
- Vitamin D2 (Active Comparator): Vitamin D2 response
  Interventions: Dietary Supplement: Vitamin D2
- Vitamin D3 (Active Comparator): Vitamin D3 response
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D + Calcium — Vitamin D 50,000 IU orally once monthly for 6 months; Calcium carbonate (as powdered limestone) 500 mg orally twice daily for 6 months
  Other Names: ergocalciferol
  Arms: Vitamin D + Calcium
Dietary Supplement: Calcium — Calcium carbonate (as powdered limestone) 500 mg orally twice daily for 6 months; Vitamin B complex (used as placebo) 1 tablet monthly for 6 months
  Other Names: limestone
  Arms: Calcium
Dietary Supplement: Vitamin D2 — 50,000 IU given orally once
  Other Names: ergocalciferol
  Arms: Vitamin D2
Dietary Supplement: Vitamin D3 — Vitamin D3 50,000 IU given orally once
  Other Names: cholecalciferol
  Arms: Vitamin D3

SUMMARY:
The purpose of this study is:

1. To compare the response of rickets to calcium with and without vitamin D.
2. To assess whether vitamin D increases calcium absorption in calcium deficiency rickets.
3. To compare the response of children with and without rickets to orally administered vitamin D3 and vitamin D2
4. To identify mutations that influence calcium and vitamin D metabolism among families of children with rickets in Nigeria and Bangladesh.
5. To assess the functional status of the 25-hydroxylase enzyme in families possessing a 25-hydroxylase mutation.

DETAILED DESCRIPTION:
Previous studies of Nigerian children with rickets demonstrated the superiority of calcium over vitamin D in producing healing. It is not known whether the addition of vitamin D to calcium will produce a better response to treatment than calcium alone in Nigerian children. A previous study suggested the possibility that vitamin D may augment the effect of calcium. We will compare the response of rickets to calcium with and without vitamin D. In addition, very little human data clearly demonstrates the effect of supplemental vitamin D on calcium absorption. We will assess whether oral vitamin D increases the already high calcium absorption even further.

Recent published data indicate that the increase in serum 25-hydroxyvitamin D may be more sustained with vitamin D3 than with vitamin D2. We will compare the response of Nigerian children with and without rickets to orally administered vitamin D3 and vitamin D2.

Because nutritional rickets tends to run in families, we will also examine amplified DNA for evidence of mutations that influence calcium and vitamin D metabolism among families of children with rickets in Nigeria and Bangladesh. Families possessing a recently identified 25-hydroxylase mutation will be given oral vitamin D2 and vitamin D3 to determine the functional status of the 25-hydroxylase enzyme.

ELIGIBILITY:
Inclusion Criteria:

* Clinical features of rickets
* Active rickets on X-ray

Exclusion Criteria:

* Treatment with calcium or vitamin D in preceding 30 days

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2004-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
XR healing of rickets | 6 months

SECONDARY OUTCOMES:
Alkaline phosphatase | 6 months
Serum calcium | 6 months
25-hydroxyvitamin D | 6 months
1,25-dihydroxyvitamin D | 2 weeks
Calcium absorption | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Thacher, MD, Principal Investigator — Mayo Clinic, Jos University Teaching Hospital
Locations (1):
- Jos University Teaching Hospital, Jos, Plateau State, Nigeria

REFERENCES:
- [Background] Thacher TD, Fischer PR, Pettifor JM, Lawson JO, Isichei CO, Reading JC, Chan GM. A comparison of calcium, vitamin D, or both for nutritional rickets in Nigerian children. N Engl J Med. 1999 Aug 19;341(8):563-8. doi: 10.1056/NEJM199908193410803. PMID 10451461
- [Background] Graff M, Thacher TD, Fischer PR, Stadler D, Pam SD, Pettifor JM, Isichei CO, Abrams SA. Calcium absorption in Nigerian children with rickets. Am J Clin Nutr. 2004 Nov;80(5):1415-21. doi: 10.1093/ajcn/80.5.1415. PMID 15531695
- [Background] Thacher TD, Fischer PR, Isichei CO, Pettifor JM. Early response to vitamin D2 in children with calcium deficiency rickets. J Pediatr. 2006 Dec;149(6):840-4. doi: 10.1016/j.jpeds.2006.08.070. PMID 17137904
- [Background] Fischer PR, Thacher TD, Pettifor JM, Jorde LB, Eccleshall TR, Feldman D. Vitamin D receptor polymorphisms and nutritional rickets in Nigerian children. J Bone Miner Res. 2000 Nov;15(11):2206-10. doi: 10.1359/jbmr.2000.15.11.2206. PMID 11092401
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Thacher TD, Fischer PR, Pettifor JM. Vitamin D treatment in calcium-deficiency rickets: a randomised controlled trial. Arch Dis Child. 2014 Sep;99(9):807-11. doi: 10.1136/archdischild-2013-305275. Epub 2014 Apr 19. PMID 24748637